CLINICAL TRIAL: NCT06686849
Title: Comparing Technological and Relational Approaches to Support Families After a Missed Well Child Visit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00118696; 1R21MD019434-01A1 (NIH)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Well-child Care Visits
Keywords: Well-Child care; Community Health Workers; Missed healthcare appointments; Text message follow-up

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care as Usual (No Intervention): In the comparison group, patients' caregivers will not be subject to any standardized follow-up procedure.
- Low-touch: Text messaging only (Experimental): The patients' primary caregiver will receive a text message that includes details about the missed appointment, and guidance on rescheduling. Up to three total reminders will be sent, spaced one week apart, if the appointment is not rescheduled in the interim.
  Interventions: Behavioral: Low-touch: texting
- High-touch: Community Health Worker outreach (Experimental): Regardless of rescheduling status, the Community Health Worker (CHW) will reach out to the primary phone number on file within approximately 1 week of enrollment in the study. Per usual team protocol, up to three phone call attempts will be made to the primary phone number on file, followed by an attempt to the secondary phone number on file. The CHW will screen the families' needs per their usual protocol and inquire about reasons for no-showing for the scheduled appointment; additional questions will include whether they can provide support for rescheduling the no-showed visit and helping to attend it. The CHW will also have a discretionary fund available through this project to help support the family in addressing instrumental needs if existing resources are not available through the hospital, governmental services, or other organizations.
  Interventions: Behavioral: High-touch: Community health worker outreach

INTERVENTIONS:
Behavioral: Low-touch: texting — Text message: The patients' primary caregiver will be sent up to three text messages spaced one week apart, starting at one week post no-show. The message will identify the child by the first name and give information about the missed visit (date, time, clinic location) and how to reschedule (by clinic-specific phone number, and/or directing the patient to myatriumhealth.org). If a patient has a newly scheduled well-child visit on file prior to all three text messages being sent, messages will be stopped.
  Arms: Low-touch: Text messaging only
Behavioral: High-touch: Community health worker outreach — Community health worker (CHW) outreach: Within approximately one week of patient enrollment and randomization to the high-touch intervention arm, the community health worker will call the primary phone number in the patient's record. Up to three phone call attempts will be made and logged for this number, then a fourth and final attempt will be made to reach the secondary contact phone number in the patient's health record. If the caregiver is successfully reached, the CHW intervention will be limited to one phone call in which the CHW will assess reason(s) why the patient missed the appointment, will screen for social and other needs, and will assist in rescheduling the missed appointment and addressing potential barriers to attendance.
  Arms: High-touch: Community Health Worker outreach

SUMMARY:
The overall goal of this study is to compare the effectiveness of different follow up protocols for scheduled but not attended ("no-show") Well-Child Visits, relative to care-as-usual (no standardized or typical follow up procedure). The main goals are to:

* Demonstrate feasibility of merging a new referral protocol following Well-Child visit no-show into existing health system Community Health Worker resources.
* Compare Well-Child Visit attendance following no-show between patients randomized to care-as-usual (comparison), text message only (low-touch intervention), and community health worker outreach (high-touch intervention) groups.
* Define the costs and cost-effectiveness of different follow-up protocols.

DETAILED DESCRIPTION:
Well-Child visits (WCV) are at the core of preventive care in pediatrics. These Visits are an important opportunity for patients to be engaged with the healthcare system, for assessing child health and development, and for screening and counseling for prevention. Missed WCVs have been associated with negative health outcomes as well as avoidable healthcare costs and may occur for a variety of different reasons. There is room for improving follow-up with families to re-engage patients after not attending a scheduled WCV ("no-show"). This study will test and compare a text messaging intervention and community health worker outreach intervention to care-as-usual (no standard follow-up) as strategies for proactively engaging families in care after no-show to promote rescheduling and visit attendance. Evaluating effectiveness and cost-effectiveness of both interventions will inform clinical practice and decision-making in healthcare to help ultimately improve pediatric preventive care.

ELIGIBILITY:
Inclusion Criteria:

* Are 0-17 years
* No-showed for a well-child visit scheduled at a family medicine or general pediatrics practice in Forsyth County, North Carolina
* Have a phone number on record for a primary caregiver
* With primary language for contact that is English or Spanish

Exclusion Criteria:

- Already rescheduled their appointment by the time the sample list was generated

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5885 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients of All Ages with any Completed Well-Child Visits | Week 6 post missed well-child visit
  Whether any Well-Child visit was completed by each patient (yes/no) following usual care, text intervention or community health worker intervention
Proportion of Patients Under 3 Years Old with any Completed Well-Child Visits | Week 6 post missed well-child visit
  Whether any Well-Child visit was completed by each patient (yes/no) following usual care, text intervention or community health worker intervention
Proportion of Patients 3 Years and Older with any Completed Well-Child Visits | Week 6 post missed well-child visit
  Whether any Well-Child visit was completed by each patient (yes/no) following usual care, text intervention or community health worker intervention
Proportion of Patients 3 Years and Older with any Completed Well-Child Visits | Month 3 post missed well-child visit
  Whether any Well-Child visit was completed by each patient (yes/no) following usual care, text intervention or community health worker intervention

SECONDARY OUTCOMES:
Proportion of Patients of All Ages with Any Rescheduled Well-Child Visit | Week 6 post missed well-child visit
  Whether any Well-Child visit was rescheduled by each patient (yes/no) following usual care, text intervention or community health worker intervention
Proportion of Patients 3 Years and Older with Any Rescheduled Well-Child Visit | Month 3 post missed well-child visit
  Whether any Well-Child visit was rescheduled by each patient (yes/no) following usual care, text intervention or community health worker intervention
Proportion of Patients of All Ages with Vaccination status up-to-date | 6 weeks post missed well-child visit
  Whether each patient is up-to-date on all age-appropriate vaccinations (yes/no)
Proportion of Patients 3 Years and Older with Vaccination status up-to-date | Month 3 post missed well-child visit
  Whether each patient is up-to-date on all age-appropriate vaccinations (yes/no)
Proportion of Patients of All Ages with Any Completed Encounter | 6 weeks post missed well-child visit
  Whether each patient had any completed healthcare encounter within the same health system (yes/no)
Proportion of Patients 3 Years and Older with Any Completed Encounter | Month 3 post missed well-child visit
  Whether each patient had any completed healthcare encounter within the same health system (yes/no)
Proportion of Patients of All Ages with Any Non-Well-Child Primary Care Visit | 6 weeks post missed well-child visit
  Whether each patient had any completed non-Well-Child primary healthcare visit within the same health system (yes/no)
Proportion of Patients 3 Years and Older with Any Non-Well-Child Visit Primary Care Visit | Month 3 post missed well-child visit
  Whether each patient had any completed non-Well-Child primary healthcare visit within the same health system (yes/no)
Proportion of Patients of All Ages with Any Specialist Visit | 6 weeks post missed well-child visit
  Whether each patient had any completed non-Well-Child specialist visit within the same health system (yes/no)
Proportion of Patients 3 Years and Older with Any Specialist Visit | Month 3 post missed well-child visit
  Whether each patient had any completed non-Well-Child specialist visit within the same health system (yes/no)
Proportion of Patients of All Ages with Any Emergency Department Visit | 6 weeks post missed well-child visit
  Whether each patient had any Emergency Department visit within the same health system (yes/no)
Proportion of Patients 3 Years and Older with Any Emergency Department Visit | Month 3 post missed well-child visit
  Whether each patient had any Emergency Department within the same health system (yes/no)
Proportion of Patients of All Ages with Any Hospitalization | 6 weeks post missed well-child visit
  Whether each patient had any hospitalization within the same health system (yes/no)
Proportion of Patients 3 Years and Older with Any Hospitalization | Month 3 post missed well-child visit
  Whether each patient had any hospitalization within the same health system (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Beata Debinski, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Department of Family and Community Medicine, Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will preserve and share predominantly transformed analytical variables, or de-identified patient data about:
  * study arm assignment
  * preferred language of care (English/Spanish)
  * prior Well-child visit in previous 2 years (yes/no)
  * age in years
  * racial categorization
  * ethnicity
  * insurance status (categorized into private, public, or uninsured)
    -# of siblings who no-showed in study period
  * unique identifier for each patient
  * unique identifier for each household
  * qualifying Well-child visit no-show encounter-level data that will be shared will be a unique identifier for the clinic location, time of visit, and a week of the year (1-52) instead of date of visit to reduce identifiability but provide information about relative time of year and season
  * dichotomized outcome data on subsequent healthcare encounters
  * dichotomized or categorized Community Health Worker-generated data (high-touch intervention group only)
Supporting Information: Study Protocol
Time Frame: Data from the first six months of trial enrollment will be deposited approximately nine months after the enrollment begins. A complete dataset for the full twelve months of enrollment will be deposited by six months after enrollment is completed. As data will be deposited to open Inter-University Consortium for Political & Social Research (openICPSR), it will be published and immediately available to the public. Data will be available on openICPSR permanently.
Access Criteria: The study protocol and codebooks (with variable-level details) will be made available as PDFs on the openICPSR website along with the data. openICPSR will also release metadata about the project that adheres to the Data Documentation Initiative (DDI) disciplinary metadata standard. The only requirements to access downloadable, de-identified data through ICPSR are user registration and agreement to ICPSR's Terms of Use, which require users to agree to not redisseminate data, to use appropriate data citation, and to maintain human subjects protections.